CLINICAL TRIAL: NCT02312739
Title: Nitrous Oxide for Pain Management During In-office Transcervical Sterilization
Acronym: NEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Society of Family Planning (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNMHSC13-594
Record Dates: First submitted 2014-10-24; First posted 2014-12-09 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-05

CONDITIONS: Contraception; Inhalation of Nitrous Oxide
Keywords: pain assessment; pain measurement; patient satisfaction; anxiety; analgesia and anesthesia; female sterilization
MeSH Terms: conditions — Patient Satisfaction; Anxiety Disorders; Agnosia | interventions — acetaminophen, hydrocodone drug combination; Lorazepam; Oxygen; Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vicodin, Lorazepam and Oxygen (Active Comparator): Patients in this group will receive the Standard Oral Pain Medications consisting of Vicodin and Lorazepam, as well as intramuscular ketorolac at least 30 minutes prior to the procedure. Oxygen via scented mask will also given.
  All participants randomized to this group will undergo in-office transcervical sterilization (Essure® procedure ) using standard technique.
  Interventions: Procedure: In-office Transcervical Sterilization (Essure®); Drug: Standard Oral pain medications; Drug: Intramuscular Ketorolac; Other: Oxygen
- Placebo pills and Nitrous Oxide (Experimental): Patients in this group will receive two placebo pills, as well as intramuscular ketorolac at least 30 minutes prior to the procedure. Nitrous oxide will be administered during the procedure via scented mask.
  All participants randomized to this group will undergo in-office transcervical sterilization (Essure® procedure ) using standard technique.
  Interventions: Procedure: In-office Transcervical Sterilization (Essure®); Drug: Intramuscular Ketorolac; Drug: Placebo pills; Other: Nitrous Oxide

INTERVENTIONS:
Procedure: In-office Transcervical Sterilization (Essure®) — The standard transcervical sterilization procedure is not being evaluated in this study, and will be performed in the same manner in the two study arms. The procedure includes a standardized paracervical block with 1% lidocaine. A 5mm operative hysteroscope is passed through the cervix and into the uterine cavity using normal saline for uterine distention. Each tubal ostium is identified, followed by deployment of the device into each fallopian tube. A confirmatory test, hysterosalpingogram, is required at 90 days post procedure to demonstrate successful sterilization.
  Other Names: Essure®; Non-surgical permanent birth control; Transcervical sterilization; Hysteroscopic sterilization
Drug: Standard Oral pain medications — one 5/325mg hydrocodone/acetaminophen (Vicodin) tablet and one 1mg Lorazepam tablet given to patients randomized to the active comparator arm at least 30 minutes before the procedure
  Other Names: Vicodin; Lorazepam
  Arms: Vicodin, Lorazepam and Oxygen
Drug: Intramuscular Ketorolac — 30mg of intramuscular ketorolac given to all patients at least 30 minutes before the procedure
  Other Names: IM ketorolac
Drug: Placebo pills — Two placebo bills given to patients randomized to the experimental arm at least 30 minutes prior to the procedure
  Other Names: Placebo
  Arms: Placebo pills and Nitrous Oxide
Other: Oxygen — Oxygen at 5L/min given to patients randomized to the active comparator arm
  Other Names: O2
  Arms: Vicodin, Lorazepam and Oxygen
Other: Nitrous Oxide — Nitrous oxide with a maximum titration of up to 70% given to patients randomized to the experimental arm
  Arms: Placebo pills and Nitrous Oxide

SUMMARY:
This is a randomized, double blind study that aims to measure the difference in maximum pain experienced during in-office transcervical sterilization (Essure®) for women receiving either inhaled nitrous oxide or standard oral analgesia (Vicodin and Lorazepam) with inhaled oxygen.

The investigators hypothesize that inhaled nitrous oxide will reduce the pain experienced more than standard oral medications in women undergoing in-office transcervical sterilization.

DETAILED DESCRIPTION:
Hysteroscopic permanent sterilization with Essure® is increasingly performed in the outpatient setting. No optimal outpatient analgesia regimen has been identified for the Essure® procedure. The investigators propose a study of inhaled nitrous oxide administered with oxygen, hereafter referred to as nitrous oxide (NO), as an intervention to lower pain experienced during the in-office procedure. The investigators hypothesize that, compared to standard oral medications, inhaled NO will decrease patient anxiety associated with the in-office procedure, as well as increase patient satisfaction and provider perceived ease of device insertion.

Women presenting to the clinic for family planning will receive our standard counseling on all forms of contraception, including short and long acting reversible contraception, and methods for permanent sterilization. Once the patient decides to have a sterilization procedure with the transcervical approach (Essure® procedure), she will undergo the standard pre-procedure evaluation, which includes a complete history, appropriate physical examination including pelvic examination, and urine pregnancy test.

Eligible women interested in sterilization will be advised of the study as an investigation evaluating nitrous oxide as an alternative to our current oral sedation pain management for in-office procedures. If they choose hysteroscopic sterilization, they will undergo informed consent for the Essure® procedure. Providers will assess patient eligibility criteria for possible enrollment into the study. If patients are eligible and choose to participate in the research study, consent for participation will be obtained. At this time patients will be randomized to treatment group based on a predetermined randomization scheme. For this research study comparing the use of NO versus oral pain medications, the NO group will receive two placebo pills and the standard group will receive one 5/325 mg oral tablet of Vicodin and one 1 mg oral tablet of lorazepam 30 minutes prior to the procedure. The standard care group will receive oxygen (instead of NO) during the procedure. All participants will receive 30 mg of intramuscular ketorolac 30 minutes prior to the procedure.

NO or oxygen will be administered via a scented nasal mask to blind patients to the intervention. NO can be titrated up to a concentration of 70% nitrous oxide and 30% oxygen based on desired analgesic effects per a predetermined sedation scale as part of the University of New Mexico Center for Reproductive Health (UNM CRH) nitrous administration protocol. All patients will be monitored with a pulse-oximeter. The patient will be fitted to their mask once the procedure is ready to begin. A single nurse will administer nitrous oxide and oxygen for all procedures. Every study patient will receive a minimum of 3 minutes of oxygen at the end of the procedure to minimize the side effects of NO. Additional oxygen will be administered as needed if a patient is experiencing residual effects of NO.

Prior to the procedure and study medications, patients will complete patient information and demographics questionnaire and will receive instruction on the 0-100mm visual analogue scale (VAS) and Spielberger State-Trait Anxiety Inventory (STAI). A baseline pain score will be recorded using the 0-100mm VAS with anchors 0 equals no pain and 100 equals worst pain imaginable, as well as baseline anxiety level using the STAI. At placement of the paracervical block and deployment of the second device coil, pain will be assessed again with the same 0-100mm VAS. At 3 to 5 minutes following completion of the procedure, maximal pain experienced during transcervical sterilization will be assessed by the patient. Prior to discharge from the clinic, the patient will rate her pain level using the same 0-100mm VAS, rate her level of anxiety with the procedure using the same STAI, and rate her overall satisfaction with the procedure measured using a 5-point Likert scale.

Immediately after the procedure, the physician will complete a 0-100mm VAS on ease of insertion of the sterilization devices with anchors 0 equals no difficulty and 100 equals very difficult. The physician will also complete a 0-100mm VAS on hysteroscopic procedure difficulty with anchors 0 equals no difficulty and 100 equals very difficult.

The standard transcervical sterilization procedure is not being evaluated in this study. After patients complete the procedure, they are contacted approximately 75 days from the procedure date to schedule a confirmatory test, hysterosalpingogram, which is required at 90 days to demonstrate successful sterilization.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women desiring permanent sterilization and have chosen to proceed with a transcervical sterilization approach
* Speaks English or Spanish
* If relying on state or federal funding for sterilization, must have appropriate federal consents signed 30 days prior to the sterilization procedure
* Agrees to either a hormonal endometrial preparation prior to the procedure or schedule the procedure during the follicular phase (days 5 through 12) of their menstrual cycle
* Sexually active who agrees to contraception for 3 months post procedure, including condoms, followed by a hysterosalpingogram (HSG) for confirmation of fallopian tubal occlusion.

Exclusion Criteria:

* With contraindications for nitrous oxide including: respiratory infection, chronic obstructive pulmonary disease (COPD), intoxication or use of street drugs, inability to breathe through their nose.
* Have taken narcotic pain medications prior to coming to their appointment
* Unsure about desire to end fertility
* History of pelvic inflammatory disease in the past 3 months
* Pregnancy or suspicion of pregnancy
* Delivery or termination of a pregnancy within the last 6 weeks
* Known allergy to contrast
* Uterine anomalies
* Previous tubal surgery
* Cervical or endometrial cancer
* Allergy to Vicodin, lorazepam, or lidocaine.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rameet Singh, MD, MPH, Principal Investigator — UNM OB GYN Division of Family Planning
Locations (1):
- UNM Center for Reproductive Health, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vicodin, Lorazepam and Oxygen: Patients in this group will receive the Standard Oral Pain Medications consisting of Vicodin and Lorazepam, as well as intramuscular ketorolac at least 30 minutes prior to the procedure. Oxygen via scented mask will also given.
  All participants randomized to this group will undergo in-office transcervical sterilization (Essure® procedure ) using standard technique.
  Standard Oral pain medications: one 5/325mg hydrocodone/acetaminophen (Vicodin) tablet and one 1mg Lorazepam tablet given to patients randomized to the active comparator arm at least 30 minutes before the procedure
  Intramuscular Ketorolac: 30mg of intramuscular ketorolac given to all patients at least 30 minutes before the procedure
  Oxygen: Oxygen at 5L/min given to patients randomized to the active comparator arm
- Placebo Pills and Nitrous Oxide: Patients in this group will receive two placebo pills, as well as intramuscular ketorolac at least 30 minutes prior to the procedure. Nitrous oxide will be administered during the procedure via scented mask.
  All participants randomized to this group will undergo in-office transcervical sterilization (Essure® procedure ) using standard technique.
  Intramuscular Ketorolac: 30mg of intramuscular ketorolac given to all patients at least 30 minutes before the procedure
  Placebo pills: Two placebo bills given to patients randomized to the experimental arm at least 30 minutes prior to the procedure
  Nitrous Oxide: Nitrous oxide with a maximum titration of up to 70% given to patients randomized to the experimental arm
Period: Overall Study
Arm/Group | Vicodin, Lorazepam and Oxygen | Placebo Pills and Nitrous Oxide
Started | 36 | 36
Withdrawn Prior to Procedure | 6 | 2
Completed | 30 | 34
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vicodin, Lorazepam and Oxygen | Placebo Pills and Nitrous Oxide | Total
Number analyzed (Participants) | 30 | 34 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (6.6) | 33.6 (4.9) | 34.1 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 64
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 26 | 47
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 13 | 9 | 22
  Hispanic/Mexican/Spanish | 14 | 16 | 30
  Native American/Alaska native | 0 | 3 | 3
  More than one | 1 | 1 | 2
  Unknown | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 30 | 34 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Scale Measurement During and After the Procedure
Description: Pain is assessed using a 0-100mm VAS with anchors 0 equals no pain and 100 equals worst pain imaginable. It is taken at baseline, after paracervical block injection and after placement of second Essure® coil. A final pain assessment is done prior to discharge.
Time Frame: At baseline before the procedure, during the procedure after paracervical block injection and after placement of second Essure® coil, and prior to discharge from clinic (approximately 30-45 minutes postprocedure)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin, Lorazepam and Oxygen | Placebo Pills and Nitrous Oxide
Number analyzed (Participants) | 30 | 34
units on a scale
  Baseline Pain | 1.1 (3.2) | 2.5 (6.7)
  After Parcervical Block | 15.6 (22.2) | 15.4 (24.3)
  At Second Coil Placement | 40.7 (33.5) | 14.9 (23.6)
  Pain at Clinic Discharge | 20.4 (21.9) | 12.4 (15.8)

2. Primary Outcome: Pain Scale Measurement - Maximum Pain Experienced
Description: The maximum pain that was experienced during the procedure is assessed using a 0-100mm VAS with anchors 0 equals no pain and 100 equals worst pain imaginable. It is taken at 3 to 5 minutes following completion of the procedure.
Time Frame: At 3-5 minutes after the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin, Lorazepam and Oxygen | Placebo Pills and Nitrous Oxide
Number analyzed (Participants) | 30 | 34
units on a scale | 54.5 (32.7) | 22.8 (27.6)

3. Secondary Outcome: Change From Baseline in Patient Anxiety Scale After the Procedure
Description: Participants were asked to complete a validated short form of the Spielberger State-Trait Anxiety Inventory (STAI) at baseline and at 3-5 minutes after the in-office sterilization procedure. On the STAI scale, participants rated five statements (I feel calm, I am tense, I feel upset, I am relaxed, I am worried) on a 1 - 4 scale (Not at all, Somewhat, Moderately, Very Much, totaling in a score from 0-20 (0 being least anxious, 20 being the most anxious).
Time Frame: At baseline before the procedure and at 3-5 minutes after the Essure® procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin, Lorazepam and Oxygen | Placebo Pills and Nitrous Oxide
Number analyzed (Participants) | 30 | 34
units on a scale
  Pre-procedure | 8.4 (2.7) | 9.4 (2.9)
  Post-procedure | 8.5 (2.9) | 8.2 (2.8)

4. Secondary Outcome: Patient Satisfaction (5-point Likert Scale)
Description: Patients were asked to rate their overall satisfaction with the procedure using a 5-point Likert scale (Very unsatisfied, Unsatisfied, Neutral, Satisfied, Very satisfied). Results were analyzed to portray the percentage of participants who felt satisfied at the listed interval levels.
Time Frame: Prior to discharge from clinic, approximately 30-45 minutes post-procedure
Measure: Number; unit: percentage of participants
Arm/Group | Vicodin, Lorazepam and Oxygen | Placebo Pills and Nitrous Oxide
Number analyzed (Participants) | 30 | 34
percentage of participants
  Very satisfied/satisfied with pain management | 77 | 85
  Neutral, unsatisfied or very unsatisfied | 23 | 15

5. Secondary Outcome: Provider Ease of Insertion (0-100mm VAS)
Description: Physician who did the procedure will complete a 0-100mm VAS on ease of insertion of the sterilization devices with anchors 0 equals no difficulty and 100 equals very difficult.
Time Frame: Within 5 minutes after the Essure® procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin, Lorazepam and Oxygen | Placebo Pills and Nitrous Oxide
Number analyzed (Participants) | 30 | 34
units on a scale | 22.7 (24.8) | 19.8 (20.7)

ADVERSE EVENTS:
Arm/Group | Vicodin, Lorazepam and Oxygen | Placebo Pills and Nitrous Oxide
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/34
Other Adverse Events (participants affected / at risk) | 0/30 | 0/34

LIMITATIONS AND CAVEATS:
Limitations of the study include the limited ability to truly blind physicians due to the signs and symptoms of N2O/O2 sedation being apparent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No